CLINICAL TRIAL: NCT01499173
Title: A Community Partnership to Treat Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Lesli E. Skolarus, MD, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GRANT10624910; 1K23NS073685-01 (NIH)
Record Dates: First submitted 2011-12-14; First posted 2011-12-26 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke preparedness intervention (Experimental): Youth and adults from predominately African American churches in Flint will be enrolled to undergo a faith-based, scientific theory-driven, peer-led behavioral intervention utilizing a pre-post test design.
  Interventions: Behavioral: Stroke Preparedness Intervention

INTERVENTIONS:
Behavioral: Stroke Preparedness Intervention — A faith-based, scientific theory-driven, peer-led behavioral intervention performed in a group setting in African American churches.

SUMMARY:
Getting to the hospital quickly is the key to treating stroke. African Americans suffer more strokes with worse outcomes and receive stroke treatments less often than European Americans. This project will work to reduce these health disparities by creating and testing the feasibility of a peer-led faith-based behavioral intervention in an African American community with a goal to increase calls to 911 so stroke patients can be treated quickly.

ELIGIBILITY:
Inclusion Criteria:

To meet participant eligibility criteria, individuals must be 18 years of age or older (adult intervention) or between 10-17 years of age (youth intervention), a resident of the Flint or greater Flint community, and English speaking.

Exclusion Criteria:

We will attempt to exclude those who cannot read English because they will not be able to benefit from the intervention materials. These criteria will be confirmed during assessment procedures prior to enrollment.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesli Skolarus, MD, Principal Investigator — University of Michigan
Locations (1):
- Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skolarus LE, Zimmerman MA, Bailey S, Dome M, Murphy JB, Kobrossi C, Dombrowski SU, Burke JF, Morgenstern LB. Stroke Ready Intervention: Community Engagement to Decrease Prehospital Delay. J Am Heart Assoc. 2016 May 20;5(5):e003331. doi: 10.1161/JAHA.116.003331. PMID 27208000

RESULTS

PARTICIPANT FLOW:
Groups:
- Stroke Preparedness Intervention: Youth and adults from predominately African American chruches in Flint will be enrolled to undergo a faith-based, scientific theory-driven, peer-led behavioral intervention utilizing a pre-post test design.
  Stroke Preparedness Intervention: A faith-based, scientific theory-driven, peer-led behavioral intervention performed in a group setting in African American churches.
Period: Overall Study
Arm/Group | Stroke Preparedness Intervention
Started | 101
Completed | 64
Not Completed | 37

BASELINE CHARACTERISTICS:
Arm/Group | Stroke Preparedness Intervention
Number analyzed (Participants) | 101
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: we present the age of the youth and adults separately
  years
    adults: number analyzed (Participants) | 73
    adults | 56 [35 to 65]
    youth: number analyzed (Participants) | 28
    youth | 14 [11 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 101
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: Completion
Description: Number of participants who complete the intervention
Time Frame: 1 week
Population: descriptive
Measure: Count of Participants; unit: Participants
Arm/Group | Stroke Preparedness Intervention
Number analyzed (Participants) | 101
Participants | 64

2. Secondary Outcome: Mean Change in Behavioral Intent to Call 911
Description: The pre-test is conducted one week prior to the post-test. A higher score indicates greater behavioral intent. Behavioral intent is measured on a scale of 0 - 8, where 0 indicates no correct answers in responses to scenarios, and 8 indicates appropriate responses (calling 911 every time it is appropriate) to the scenarios presented.
Time Frame: 1 week elapsed between a pretest before 1st workshop and post-test at the end of 2nd workshop
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Stroke Preparedness Intervention
Number analyzed (Participants) | 64
units on a scale
  pre-test | 4.4 [4.2 to 4.6]
  post-test | 5.2 [4.9 to 5.5]
Statistical Analysis 1: Comparison: Stroke Preparedness Intervention; Test type: Superiority; p < 0.01, multilevel linear regression — Actual p value shown here; not threshold

3. Secondary Outcome: Mean Change in Stroke Recognition
Description: Stroke recognition was scored on a 0 - 9 point scale where 0 represents no correct answers regarding 9 scenarios and 9 represents perfect stroke recognition.
Time Frame: 1 week elapsed between a pretest before 1st workshop and post-test at the end of 2nd workshop
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Stroke Preparedness Intervention
Number analyzed (Participants) | 64
units on a scale
  pre-test | 5.9 [5.6 to 6.1]
  post-test | 6.0 [5.7 to 6.3]
Statistical Analysis 1: Comparison: Stroke Preparedness Intervention; Test type: Superiority; p = 0.34, multilevel linear regression

4. Secondary Outcome: Perception of Social Norms Clustered Within Churches Across Multiple Time Points
Description: Perception of social norms is measured by the odds ratio of the responses to questions of participant agreement with others' influence to calling 911 if he/she were to see a stroke. Odds ratios measure the odds of responses, so higher odds ratios suggest greater odds of the positive change in social norms in the post-test compared to the pre-test. Questions: 1) Most people would call 911 if they were to see a stroke. 2) My family would want me to call 911 if I were to see a stroke. Given that participants within each church are more alike than participants between churches and the multiple time points, hierarchical models were used. Specifically, multilevel mixed-effects ordered logistic regression models with a fixed church-level intercept and a random participant level intercept were used to explore change between baseline and immediate post-test and baseline and delayed post-test social norms after accounting for the participants' church.
Time Frame: 1 week between pretest before 1st workshop and post-test at the end of 2nd workshop and 1 month till the delayed post test
Measure: Number; unit: odds ratio
Arm/Group | Stroke Preparedness Intervention
Number analyzed (Participants) | 64
odds ratio
  1 wk: Q1: Most people would call 911 | -0.5
  1 wk: Q2: My family would want me to call 911 | 0.2
  1 mo: Q1: Most people would call 911 | -0.9
  1 mo: Q2: My family would want me to call 911 | 0.1
Statistical Analysis 1: Comparison: Stroke Preparedness Intervention; Odds ratio was calculated for each question comparing 1 week data with 1 month data; Test type: Other — odds ratio; Odds Ratio (OR) = -0.5

5. Secondary Outcome: Perception of Self-efficacy Clustered Within Churches Across Multiple Time Points
Description: Perception of self-efficacy is measured by the odds ratios of the responses to questions of participant confidence in being able to identify and respond appropriately to a stroke. Odds ratios measure the odds of responses, so higher odds ratios suggest greater odds of positive self-efficacy change in the post-test compared to the pretest. Questions asking about self-efficacy were:1) I would be able to tell if someone is having a stroke and 2) I know what to do if I saw someone having a stroke. Given that participants within each church are more alike than participants between churches and multiple time points hierarchical models were used. Specifically, multilevel mixed-effects ordered logistic regression models with a fixed church-level intercept and a random participant level intercept were used to explore change between baseline and immediate post-test and baseline and delayed posttest self-efficacy after accounting for the participants' church.
Time Frame: as for outcome 4
Measure: Number; unit: odds ratio
Arm/Group | Stroke Preparedness Intervention
Number analyzed (Participants) | 64
odds ratio
  1 wk: Q 1: I'd be able to tell | 1.2
  1 wk: Q2: I know what to do | .8
  1 mo. Q 1: I'd be able to tell | .8
  1 mo: Q2: I know what to do | .3

6. Secondary Outcome: Perception of Stroke Attitude Clustered Within Churches Across Multiple Time Points
Description: Stroke attitude is measured by the odds ratio of participant's positive perception of calling 911 for stroke. Odds ratios measure the odds of responses, so higher odds ratios suggest greater odds of stroke attitude change in the post-test compared to pre-test. Stroke attitude questioners were: Q1) If I were to see signs of a stroke, calling 911 would be... (range "extremely pleasant" to "very unpleasant); and Q2) If a person has signs of a stroke, calling 911 right away could be... (range "very helpful" to "very harmful). Given that participants within each church are more alike than participants between churches and multiple time points, hierarchical models were used. Specifically, multilevel mixed-effects ordered logistic regression models with a fixed church-level intercept and a random participant level intercept were used to explore change between baseline and immediate post-test and baseline and delayed post-test stroke attitude after accounting for the participants' church.
Time Frame: as for outcome 4
Measure: Number; unit: Odds ratio
Arm/Group | Stroke Preparedness Intervention
Number analyzed (Participants) | 64
Odds ratio
  1 wk: Q1: If I were to see... | .05
  1 wk: Q2: If a person has signs of a stroke... | 0.3
  1 mo: Q1: If I were to see... | -0.07
  1 mo: Q2: If a person has signs of a stroke... | -0.5

7. Other Pre Specified Outcome: Program Satisfaction
Description: Program satisfaction is measured by percentage of participants that completed the program who answered on the post test: very satisfied or extremely satisfied on a questionnaire about the program.
Time Frame: 1 week elapsed between a pretest before 1st workshop and post-test at the end of 2nd workshop
Measure: Number; unit: percentage of participants
Arm/Group | Stroke Preparedness Intervention
Number analyzed (Participants) | 64
percentage of participants | 80

ADVERSE EVENTS:
Arm/Group | Stroke Preparedness Intervention
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 0/101

LIMITATIONS AND CAVEATS:
Because this was a pre-post design, it cannot be the basis for a conclusion that Stroke Ready caused an increase in stroke preparedness and psychological variables

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No